CLINICAL TRIAL: NCT01191658
Title: Can Neck Circumference Measurements Less Than 43cm or Greater Than 43cm Predict Difficulty of Tracheal Intubation?
Status: Completed | Type: Observational
Sponsor: CAMC Health System (Other)
Responsible Party: William White, Jr., DMP, CRNA, CAMC Institute
Other Study IDs: 10-07-2252
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Neck Circumference, Difficulty of Tracheal Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The circumference of a person's neck is a useful predictor of difficulty of insertion of a breathing tube.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1-4
* Receiving general endotracheal anesthesia for surgery

Exclusion Criteria:

* Limited range of motion of the neck or jaw
* Cervical spine injuries
* Upper airway pathology
* Previous facial trauma, or goiter
* Patients receiving regional anesthesia or anesthesia other than general, endotracheal anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients who require tracheal intubation for general anesthesia and surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States